CLINICAL TRIAL: NCT01224457
Title: Effect of CYP2C9/CYP2C19 Polymorphism on Pharmacokinetics of Phenobarbital in Korean Neonatal Seizure Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 4-2008-0029
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Neonatal Seizure
MeSH Terms: interventions — Phenobarbital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Phenobarbital — phenobarbital 20mg/kg iv infusion, after 24hours of loading, 2.5mg/kg bid daily

SUMMARY:
The pharmacogenomic profiles of drug metabolizing enzymes play an important role in pharmacokinetics (PK) of drugs. Phenobarbital (PB), worldwidely used for neonatal seizure, is a drug that requires careful dose adjustments based on therapeutic drug monitoring. It was reported that phenobarbital (PB) metabolism was affected by CYP2C9 and CYP2C19 polymorphisms in adults. This study aims to evaluate the effects of the CYP2C9 and CYP2C19 genetic polymorphisms on PB PK in infants with neonatal seizure for an optimal dosing strategy.

ELIGIBILITY:
Inclusion Criteria:

* Infant treated by phenobarbital monotherapy, diagnosed neonatal seizure
* Infant taken the drug concentration one more time
* given the informed consent

Exclusion Criteria:

* progressed CNS disorder
* severe systemic illness
* GOT/GPT level more than 2times of normal value,more than 3times elevation of BUN/creatinine level
* congenital hemolytic anemia
* genetic disorder

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
pb drug concentration | 48 hours after administering phenobarbital
  pb drug concentration, CYP2C9/CYP2C19 polymorphism